CLINICAL TRIAL: NCT04991467
Title: A Multimodal Parent-focused Intervention for Vulnerable Populations in the Bronx
Acronym: CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Miami (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2020-12561; R01MH126821 (NIH)
Record Dates: First submitted 2021-07-16; First posted 2021-08-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Parenting; Covid19
Keywords: COVID; Parental Stress; Social Determinants of Health; Valera
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: 3 interventions: Care & Valera, Care only, and Valera only.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Parents of children receiving mental health treatment at Montefiore (Experimental): Participants will either CARE program alone; b) Valera Health app; c) CARE program and Valera Health app .
  Interventions: Behavioral: CARE Program and Valera Application with care manager functionality; Behavioral: Valera Application with care manager functionality; Behavioral: CARE Program
- Parents of children being treated for autoimmune disorders at Montefiore (Experimental): Participants will either CARE program alone; b) Valera Health app; c) CARE program and Valera Health app.
  Interventions: Behavioral: CARE Program and Valera Application with care manager functionality; Behavioral: Valera Application with care manager functionality; Behavioral: CARE Program
- Healthcare workers at Montefiore (Experimental): Participants will either CARE program alone; b) Valera Health app; c) CARE program and Valera Health app.
  Interventions: Behavioral: CARE Program; Behavioral: Valera Application; Behavioral: CARE Program and Valera Application

INTERVENTIONS:
Behavioral: CARE Program and Valera Application with care manager functionality — Participant will take part in 12 week CARE program and receive the Valera health application which will provide parent education materials as well as the ability to connect to their child's treatment team via care manager.
  Arms: Parents of children being treated for autoimmune disorders at Montefiore; Parents of children receiving mental health treatment at Montefiore
Behavioral: Valera Application with care manager functionality — Participant will receive the Valera health application which will provide parent education materials and the ability to connect to their child's treatment team via care manger.
  Arms: Parents of children being treated for autoimmune disorders at Montefiore; Parents of children receiving mental health treatment at Montefiore
Behavioral: CARE Program — Participant will take part in 12 week CARE program.
Behavioral: Valera Application — Participant will receive the Valera health application which will provide parent education materials.
  Arms: Healthcare workers at Montefiore
Behavioral: CARE Program and Valera Application — Participant will take part in 12 week CARE program and receive the Valera health application which will provide parent education materials.
  Arms: Healthcare workers at Montefiore

SUMMARY:
For caregivers in the Bronx, the pandemic has caused unprecedented psychological distress; in addition to combating social determinants of health (SDOH), these families now face greater financial insecurity and challenges related to their school-aged children. Furthermore, social distancing requirements and limited telehealth resources for Bronx families have posed greater barriers to healthcare. Such parental distress contributes to heightened risk of transgenerational cycles of psychological stress, trauma and maltreatment. The social and economic impacts of the COVID-19 pandemic have had significant consequences for family well-being, putting parents at higher risk of experiencing distress and potentially impairing their ability to provide supportive care to their children. Although children may be less susceptible to the most damaging physical consequences of COVID-19, there are growing concerns regarding the short-and long-term impacts of pandemic-related stressors on children. The marked upheaval of family life over an extended period may make children vulnerable to mental health consequences associated with the public health crisis and infection mitigation efforts. School and childcare closures, unstable financial circumstances, social isolation and lack of support have a disproportionate, cumulative impact on parents and may undermine their capacities to provide support for their children. Importantly, a large body of evidence suggests that parental stress during times of disasters induces psychopathologies in family members including children. Further, high anxiety and depressive symptoms in parents during the pandemic have been associated with higher child abuse potential, whereas greater parental support was associated with lower perceived stress and child abuse potential. In addition to psychological impacts, stress associated with caregiving can interfere with parents' ability to maintain their own health. This multimodal study addresses key strategies to mitigate the psychological and health impact of COVID-19 in parents.

DETAILED DESCRIPTION:
Study Design

1. Objectives The study team hypothesizes that both the CARE program and the Valera Health app will mitigate the psychological effects of COVID-19 while enhancing access to healthcare in the Bronx. The study will take place at Montefiore Medical Center (MMC), the largest health system in the Bronx, serving predominantly racial and ethnic minority individuals from underserved families. This study will focus on three vulnerable caregiver cohorts presenting with moderate stress: a) caregivers of children with psychiatric conditions (N=130); b) caregivers of children with autoimmune illnesses (N=130); c) caregivers who are frontline healthcare workers at MMC (N=130). While the latter may have more favorable SDOH than families treated at MMC, this cohort has faced unprecedented stress during the pandemic. A randomized controlled trial (RCT) (Stage III, NIH model) with 3 arms will test the study hypothesis: a) CARE program alone; b) Valera Health app; and c) CARE program and Valera Health app. Study procedures will include phone screen to assess eligibility, and surveys at four timepoints: (at study enrollment, 6-, 12- and 24-weeks) will assess parental stress, reflective functioning (RF), barriers to access to healthcare, mood and anxiety symptoms, suicidality (safety) and additional parent and child clinical measures. Smartphones and connectivity will be provided as needed.

   Aim 1. To examine the efficacy of the 12-week CARE program on caregivers' emotional health and RF. Hyp. 1: (a) Compared to the Valera Health app arm at 12- and 24-week follow-up, participation in the CARE program will result in decreased caregiver's perceived stress, increased RF, and improved caregiver's mood and anxiety symptoms. (b) Therapeutic improvements in Hypothesis 1a will be mediated by RF, as it reflects mentalizing capacity.

   Aim 2: To examine the efficacy of the 12-week Valera Health app on caregivers' emotional health and access to healthcare. Hypothesis 2: (a), The Valera Health app, will result in decreased caregiver's perceived stress, increased access to healthcare, and increased adherence to and engagement in treatment. (b) CARE program + Valera Health app arm will be superior to CARE or Valera Health app alone on all outcome measures.

   Exploratory Aim: (a) The study will also explore the effects on outcome of providing technology and connectivity to families who lack them during the study period. (b) The relative effectiveness of the intervention among the 3 vulnerable cohorts will be explored. (c) Machine learning approaches to explore complex patterns as predictors of outcome including COVID-19 illness/deaths, medical comorbidity, psychopathology, housing, poverty, children's school status, age, family functioning, and trauma, will be utilized.
2. Study Timelines

Individual Subject Timeline:

Participation in this research will last about 24 weeks. Participants will partake in 12 one-hour group sessions that meet once per week. Participants will complete several surveys when enrolled in the study and then after 6 weeks, after 12 weeks, and after 24 weeks.

Overall Timeline:

Because Investigators intend to rely on a pre-existing clinical infrastructure, Investigators anticipate being able to begin enrollment within the first six months of the study. Participants will return for 6-month follow-ups. Data analysis will occur throughout the duration of the study, along with publications and conference presentations. The likelihood that this study will be carried out as planned is very high, as all methods and collaborations are already in place.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be primary caregivers who present with moderate level of stress by meeting a severity score of ≥ 14 on the Perceived Stress Scale (PSS)
* Investigators will allow primary caregivers (e.g., grandmothers and aunts) as it is common in the patient population
* Clinical cohorts will be active patients in the psychiatric and rheumatology clinics in Montefiore Medical Center (MMC)
* Frontline health care providers will be those who are required to work on site at Montefiore Medical Center (MMC)

Exclusion Criteria:

* Serious psychiatric or substance use difficulty that, in the judgement of the PI, would preclude meaningful participation in a parent intervention
* Active child abuse/maltreatment cases
* Neurocognitive conditions that may prevent participants from accessing telehealth services
* Primary language other than Spanish or English
* Use of the Valera Health app or a smartphone health platform similar to the Valera app

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2021-12-17 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Caregiver Perceived Stress | From Week 0 to Week 6, Week 12, and Week 24
  Change in Caregiver Perceived Stress will be assessed using the Perceived Stress Scale (PSS). The PSS is 10-item scale which measures the degree to which situations in one's life are appraised as stressful and serves as an assessment of overall stress. Participants provide responses on the PSS based on their perceptions of stress over the prior month. Items are scored on a 5-point Likert scale ranging from 0 ("Never") to 4 ("Very Often"), for an overall possible score of 0-40. Responses to the 4 positively worded items on the scale (Items 4, 5, 7, and 8) are reverse scored (e.g., 0=4 and 4=0). Higher overall scores are associated with greater perceived stress over the past month. For purposes of this study change from baseline will be assessed and positive scores are associated with increased perceptions of stress. Scores will be summarized by study arm using basic descriptive statistics. Paired t-tests will be used to compare parental stress vs. baseline within each arm.

SECONDARY OUTCOMES:
Change in Parental Reflective Functioning (PRF) - Children | From Week 0 to Week 6, Week 12, and Week 24
  Change in PRF, for parents of children <12 years of age, will be assessed using the Parental Reflective Functioning Questionnaire (PRFQ). The PRFQ is an 18-item self-report measure designed to assess PRF or mentalizing, or the capacity to understand oneself and others in terms of mental states (e.g., feelings, desires, goals). Parents answer each item based on the extent to which they agree or disagree with the statement. Items are scored on a 7-point Likert scale ranging from 0 ("Strongly Disagree") to 7 ("Strongly Agree"), for an overall possible score of 18-126. Responses to Items 11 and 18 are reverse scored (e.g., 1=7 and 7=1). Higher overall scores are indicative of better reflective functioning. For purposes of this study change from baseline will be assessed and positive scores are associated with improved reflective functioning or mentalizing. Scores will be summarized by study arm. Paired t-tests will be used to compare reflective functioning vs. baseline within each arm.
Change in Parent Reflective Functioning (PRF) - Adolescent | From Week 0 to Week 6, Week 12, and Week 24
  Change in PRF, for parents of children >=12 years of age, will be assessed using the Parental Reflective Functioning Questionnaire for Adolescents (PRFQ-A). The PRFQ-A is an 18-item specialized version of the PRFQ tailored for parents of adolescents. Parents provide responses for each item based on the extent to which they agree or disagree with the statement. Items are scored on a 7-point Likert scale ranging from 0 ("Strongly Disagree") to 7 ("Strongly Agree"), for an overall possible score of 18-126. Responses to Items 11 and 18 are reverse scored (e.g., 1=7 and 7=1). Higher overall scores are indicative of better reflective functioning. For purposes of this study change from baseline will be assessed and positive scores are associated with improved reflective functioning or mentalizing. Scores will be summarized by study arm. Paired t-tests will be used to compare reflective functioning vs. baseline within each arm.
Change in Access to Healthcare | From Week 0 to Week 6, Week 12, and Week 24
  Change in Access to Healthcare will be assessed using the Barriers to Care Questionnaire (BCQ). The BCQ is a 39-item questionnaire designed to assess barriers to healthcare access and quality. The BCQ explores 5 domains: pragmatics, skills, marginalization, expectations, and knowledge/beliefs and helps identify factors that may prevent or delay access to healthcare. Parents are presented with a set of items and asked how much of an issue each is in getting healthcare for their children. Response options are 100 for "No Problem," 75 for "Almost Never," 50 for "Sometimes," 25 for "Often," and 0 for "Almost Always," such that higher scores reflect more positive healthcare experiences and fewer barriers to access. Overall scores are averaged. For this study change from baseline will be assessed such that positive scores are associated with fewer barriers to access. Scores will be summarized by study arm. Paired t-tests will be used to compare access scores vs. baseline within each arm.
Change in Depression | From Week 0 to Week 6, Week 12, and Week 24
  Change in depressive symptoms will be assessed using Beck's Depression Inventory (BDI). The BDI is a 21-item, self-report rating inventory that measures characteristic attitudes and symptoms of depression over time. Participants are presented with a list of statements and for each item and select the statement that best reflects their mood. Each item is rated on a 4-point Likert scale ranging from 0-3, yielding an overall possible score of 0-63. Higher overall scores are associated with greater symptom severity. For purposes of this study change from baseline will be assessed such that positive scores are associated with greater severity of depressive symptoms. Scores will be summarized by study arm using basic descriptive statistics. Paired t-tests will be used to compare parental stress vs. baseline within each arm.
Change in Anxiety | From Week 0 to Week 12, and Week 24
  Change in anxiety symptoms will be assessed using the Beck Anxiety Inventory (BAI). The BAI is a 21-item, self-report measure of severity of anxiety over the past month. Participants are presented with a list of common symptoms of anxiety and rate each set of statements on a 4-point Likert scale ranging from 0 ("Not at all") to 3 ("Severely, it bothered me a lot"), yielding an overall possible score of 0-63. Higher overall scores are associated with greater perceived severity. For purposes of this study change from baseline will be assessed such that positive scores are associated with increased perception of anxiety symptoms. Scores will be summarized by study arm using basic descriptive statistics. Paired t-tests will be used to compare parental anxiety vs. baseline within each arm.
Change in Suicidal Ideation (Safety Measure) | From Week 0 to Week 6, Week 12 and Week 24
  Change in Suicidal Ideation will be assessed using the Beck Scale for Suicidal Ideation (BSSI). The BSSI is a 19-item, self-reporting scale that measures the presence and intensity of suicidal ideation over the last week. Participants select a statement from each group of statements on the BSSI to describe how they have been feeling over the prior week. Response items are rated on an ordinal scale ranging from 0-2, yielding an overall possible score of 0-38. Higher scores reflect greater suicide risk. For purposes of this study change from baseline will be assessed and positive scores are associated with increased suicidal risk. Scores will be summarized by study arm using basic descriptive statistics. Paired t-tests will be used to compare parental suicide risk vs. baseline within each arm.

OTHER OUTCOMES:
Change in Five Minute Speech Sample | From Week 0 to Week 6, Week 12, and Week 24
  The Five Minute Speech Sample (FMSS) will be used to assess parents' expressed emotion (EE) regarding their child. Parents will call into a Montefiore phone line and will be prompted to state their name and answer 4 questions on the REDCap database screen.
Change in Multidimensional Scale of Perceived Social Support | From Week 0 to Week 24
  MSPSS
Change in Youth Outcome Questionnaire | From Week 0 to Week 24
  YOQ
Change in COVID Impact Scale | From Week 0 to Week 12 and Week 24
  COVID Impact Scale
Change in Kansas Parental Satisfaction Scale | From Week 0 to Week 6, Week 12 and Week 24
  KPSS
Change in Family Assessment Device-General Functioning Scale | From Week 0 to Week 12 and Week 24
  FAD
Change in Life Events Checklist | From Week 0 to Week 12 and Week 24
  LEC
Change in Health Related Quality of Life | From Week 0 to Week 24
  Caregiver Quality of Life
Change in PC-PTSD COVID | From Week 0 to Week 24
  PC-PTSD COVID
RaLES-B | Week 0
  Discrimination
Change in Multidimensional assessment of emotion regulation and dysregulation | From Week 0 to Week 12 and Week 24
  DERS-18
Change in Multidimensional Scale of Perceived Social Support | From Week 0 to Week 12
  MPSS
Change in PROMIS EARLY CHILDHOOD | From Week 0 to Week 24
  PROMIS EARLY CHILDHOOD
Change in PROMIS Parent Proxy Scale | From Week 0 to Week 24
  PROMIS Parent Proxy Scale
Philadelphia ACE | Week 0
  Philadelphia ACE
Change in Multidimensional Assessment of Parenting Scale (MAPS) | From Week 0 to Week 12 and Week 24
  (MAPS)
Change in Drug Abuse Screening Test | From Week 0 to Week 12 and Week 24
  DAST
Change in Alcohol Use Disorders Identification Test (Audit C) | From Week 0 to Week 12 and Week 24
  Audit C
Change in Treatment and Health Behavior Questionnaire | From Week 0 to Week 6, Week 12 and Week 24
  Treatment and Health Behavior Questionnaire
Change in Parent Stress Index | From Week 0 to Week 12 and Week 24
  PSI-4

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Alpert, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF